CLINICAL TRIAL: NCT06483438
Title: Handwriting as an Objective Tool to Support the Identification of People With Alzheimer's Disease: Suitability of an Assessment Protocol
Brief Title: Handwriting as an Objective Tool to Support the Identification of People With Alzheimer's Disease
Acronym: HAD
Status: Completed | Type: Observational
Sponsor: University of Évora (Other)
Collaborators: NOVA Medical School (Other); Faculdade de Motricidade Humana (Other); University of Lisbon (Other)
Responsible Party: Principal Investigator, Ana Rita Matias, Researcher and Assistant Professor, University of Évora
Other Study IDs: CHRC2022Handwriting&Dementia
Record Dates: First submitted 2024-06-07; First posted 2024-07-03 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-06

CONDITIONS: Dementia
Keywords: Prevention; Electroencephalography; Handwriting; Movement
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: subjects with dementia Group 2: subjects without dementia o Group/Cohort Description [*]: Group 1: subjects over the age of 50, with a diagnosis of dementia according to DSM-5 criteria and proven by neuropsychological assessment.
  Group 2: subjects over the age of 50, with no cognitive impairment on the neuropsychological assessment and with no previous neurological and/or psychiatric history or other illnesses that could interfere with the collection of writing data.

SUMMARY:
Alzheimer's disease (AD) is the most common of dementia, and has associated cognitive and motor disorders, with consequences on daily activities, including handwriting.

Handwriting has been used to study fine motor control or executive functioning in healthy and unhealthy populations. Changes in this skill are present at different stages of the clinical course of Alzheimer's Disease. The sensorimotor deterioration is observed in handwriting tasks (motion kinematics, such as movement time, speed, and profiles) and brain activity rhythms.

Handwriting has been used to study fine motor control or executive functioning in healthy and unhealthy populations, and changes in this skill are present at different stages of the clinical course of dementia. From a theoretical perspective, because sensorimotor deterioration observed in handwriting tasks (motion kinematics, such as movement time, speed, and profiles).

Due to the large number of brain areas related to handwriting performance, brain electrical activity analysis can be an early indicator of brain dysfunction. Although there is a lack of validation across healthy and non-healthy populations Electroencephalogram (EEG) measures have the potential for evaluating cognitive performance.

This research aims to analyze the suitability of the handwriting assessment protocol, which can contribute to a more in-depth knowledge of this subject and potentially support early identification and treatment.

DETAILED DESCRIPTION:
The minimum sample size for this pilot study is 75 participants, which is the minimum sample size calculated by G*power (90% power, significance level 0.05) to perform the planned between-group comparisons (ANOVA), correlations (Pearson), and nonlinear analyses. Participants who agree to participate in this study will be asked to provide demographic information, such as age, Portuguese as a native language, education level, motor/physical problems, and medical problems. By underlining the social relevance of the project, the investigators anticipate that at least 80% of the invited subjects will be interested in participating in this research.

In the first phase, the request for analysis of this project by the Ethics Committee and the Scientific Council of the University of Évora was made. After approval, the entities were contacted to present the project and start contact with the participants. Then, each participant (or their legal tutor) gave informed consent, where they were aware of the confidentiality of the data collected throughout the study and that they would not be disclosed, being only used for academic purposes.

Subjects were invited to participate in three organizations: Espírito Santo Hospital of Évora (HESE) and two Residential Centers for the Elderly. Two types of participants were recruited in these organizations. At HESE, participants with a diagnosis of dementia (validated by the medical team of the Neurology Service) and some of their healthy family members (without a diagnosis). At the Residential Centre for the Elderly, participants who did not have any medical diagnosis record were subject to a neuropsychological evaluation (lasting approximately 60 minutes) to differentiate the group of participants with and without dementia (and not to define which type of dementia). All participants will take a handwriting assessment (lasting approximately 60 minutes).

The data will be analyzed using the Statistical Package for the Social Sciences [SPSS] to conduct a cross-sectional study.

For the neuropsychological assessment, the following instruments will be used:

* Semi-structured interview of neuropsychological anamnesis. This interview was conducted directly with the individual, and will be divided into nine topics: i) personal data, ii) reason for the request, iii) clinical history, iv) school and professional background, v) complaints, vi) impact of brain injury, vii) other information, viii) the rationale of the neuropsychological assessment and ix) inventory on the anamnesis as the first occasion of evaluation (via direct observation method);
* The Geriatric Depression Scale (GDS) is a scale specifically developed for use in the elderly population, which combines administration and an easy-to-use response format. It consists of 30 items that have two possible answers (Yes; No) with two domains: cognitive and affective. The total result varies between 0 and 30 points: 0-10 points (absence of depressive symptoms),11-20 points (mild depressive symptoms) or 21-30 points (severe depressive symptoms);
* -The Mini-Mental State Examination (MMSE) is one of the most widely used instruments in screening cognitive deficits. The cut-off points are 22 for literacy from 0 to 2 years, 24 for literacy from 3 to 6 years, and 27 for literacy equal to or greater than 7 years.
* The Mattis Dementia Rating Scale (DRS-2) is a validated neuropsychological battery for assessing cognition in general, including attention, initiative/perseverance, visuospatial construction, conceptualization, and memory. The cut-off point used is the tenth percentile of normative data for the Portuguese population of age and educational level;
* Clock Design Test is a neuropsychological test, often used in dementia screening.

The handwriting assessment will be carried out by a psychomotor therapist with extensive experience. The instruments will be:

* Beery Buktenica Visual-Motor Integration Development Test - 6 (VMI-6), to be the visual-motor integration, the Portuguese translation and adaptation of the This instrument are composed of three distinct tests - Visuomotor Integration Development Test, Visual Perception Development Test and Motor Coordination Development Test - evaluates visual-motor integration, visuo-perceptual skills and motor coordination, respectively.
* Adult Writing Assessment Battery (HAB). To assess pen control, writing speed, and readability in adults, a). This battery of tests includes different subtests to assess motor and writing skills used in everyday life. Each sub-test is assessed by a specific algorithm, which determines the percentage of letters and numbers that the participant can write legibly. The final evaluation is carried out on a quotation sheet. The HAB will be carried out on a Wacom digitizing platform and the data extraction will be done through the MovAlyzeR software.
* NeuroScript MovAlyzeR software (version 6.1) will be used to analyze the performance of older adults on VMI in relation to spatial, temporal, and kinematic variables of writing.
* EPOC X is a noninvasive wireless electrophysiology procedure that will be used to assess brain activity during the handwriting task (through the HAB).
* The Movsense application enables the use of portable sensors, which can be affixed to the individual's skin or clothing and collect various biomechanical data associated with arm movement.

The data will be collected individually, directly with the individual, in the classroom using a table and a chair to perform the tasks in two sessions: one for neuropsychological assessment and the other for motor assessment. This data collection will take place after the completion of the Informed Consent.

Stroke, vertical/horizontal start position, vertical/horizontal size, slant, reaction time, duration, and pen pressure will be aggregated to obtain the handwriting cinematics.

The brain activity will be measured by the calculation of the spectral density mean from theta, alpha-1and beta bands.

Handwriting legibility will be given by the total score from HAB and the visuomotor will be reported by total and partial score from the VMI-6.

ELIGIBILITY:
Dementia group

Inclusion criteria:

* Over 50 years of age
* The inclusion criteria for the dementia group are as follows: patients diagnosed with dementia according to the DSM-5 criteria and cognitive impairment proven in the neuropsychological assessment
* Portuguese native language

Exclusion criteria:

- Previous neurological history (e.g. stroke, traumatic brain injury, multiple sclerosis, among others), psychiatric history or other incapacitating illnesses that could interfere with the collection of writing data. (NOTE that neurological disease is accepted in the dementia group, but co-morbidity of previous and actual neurological diseases will be excluded) Cognitively normal group

Inclusion criteria:

* Over 50 years of age
* At least three years of schooling

Exclusion criteria:

- Presence of neurological history (e.g., stroke, traumatic brain injury, multiple sclerosis, among others), psychiatric history, or other incapacitating illnesses that could interfere with the collection of writing data.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from Municipal and Community Associations, Senior Universities and Residential Centre for the Elderly
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2023-12-02 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Stroke | Baseline
  A stroke is a series of lines or curves written in a single letter, i.e., the path traced by the pen on the paper. Traces are analyzed movements that unite a movement pattern. A movement pattern can be segmented using 2 segmentation methods: zero crossings of the velocity profile after the velocity peak or the minimum velocity after the velocity peak. This measure is obtained through the software Movalyzer, during the handwriting tasks.
Vertical/horizontal start position | Baseline
  Initial vertical/horizontal position relative to the lower limit of the digitizer area (in cm).
Vertical/horizontal size | Baseline
  Vertical vector difference between the start and end of a stroke (in cm).
Slant | Baseline
  Segment slope, which is estimated by the orientation of the line by minimizing/reducing the sum of the squares of the perpendicular distances of all pixels to the line through the gravity point (in radians).
Reaction time | Baseline
  Is the time from the start of the recording to the start of the trace (in sec).
Duration | Baseline
  Time interval between the first and last samples in a stroke/segment (in sec).
Pen pressure | Baseline
  Average pen pressure values along a stroke (N/m2).
Brain activity | Baseline
  Spectral density mean from the frequency of the three bands (theta, alpha, beta)

SECONDARY OUTCOMES:
Handwriting legibility | Baseline
  Handwriting legibility will be obtained through the Handwriting Assessment Battery's (HAB) partial score. There is no maximum or minimum. The higher the legibility percentage, the higher the number of legible letters and numbers.
Handwriting speed | Baseline
  Handwriting speed will be obtained through the Handwriting Assessment Battery's (HAB) partial score. There is no maximum or minimum. The shorter the handwriting time, the better the handwriting speed.
Visuomotor integration | Baseline
  1. Visuomotor integration will be obtained through the total score of the test Beery Buktenica - 6 (VMI-6). There is no maximum or minimum score. The higher the raw score, the higher the percentile, which corresponds to better visuomotor integration.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Matias, PhD, Principal Investigator — University of Évora
Locations (3):
- Portugal (3):
  - Espírito Santo Hospital of Évora, Evora
  - Casa dos Avós Residence, Ponte de Sôr
  - Costa Azul Residence, Sesimbra

IPD SHARING:
Plan to Share IPD: Yes
Yes: There is a plan to make IPD and related data dictionaries available. All IPD that underlie results in a publication will be shared. Specifically, data from variables mentioned previously, age, gender, and group label.
Supporting Information: Study Protocol
Time Frame: Starting 6 months after publication
Access Criteria: Researchers who wish to have access to IPD, should contact principal researcher. The request should be done by email, were researchers should indicate: complete name, affiliation, position, and justify their interest. After the request will be evaluated by two of the elements of the research group.

REFERENCES:
- [Background] Yan JH, Rountree S, Massman P, Doody RS, Li H. Alzheimer's disease and mild cognitive impairment deteriorate fine movement control. J Psychiatr Res. 2008 Oct;42(14):1203-12. doi: 10.1016/j.jpsychires.2008.01.006. Epub 2008 Feb 15. PMID 18280503
- [Background] Stergiou N, Harbourne R, Cavanaugh J. Optimal movement variability: a new theoretical perspective for neurologic physical therapy. J Neurol Phys Ther. 2006 Sep;30(3):120-9. doi: 10.1097/01.npt.0000281949.48193.d9. PMID 17029655
- [Background] Palmis S, Danna J, Velay JL, Longcamp M. Motor control of handwriting in the developing brain: A review. Cogn Neuropsychol. 2017 May-Jun;34(3-4):187-204. doi: 10.1080/02643294.2017.1367654. Epub 2017 Sep 11. PMID 28891745
- [Background] Morgado J, Rocha CS, Maruta C, Guerreiro M, Martins IP. Cut-off scores in MMSE: a moving target? Eur J Neurol. 2010 May;17(5):692-5. doi: 10.1111/j.1468-1331.2009.02907.x. Epub 2009 Dec 29. PMID 20050900
- [Background] Harbourne RT, Stergiou N. Movement variability and the use of nonlinear tools: principles to guide physical therapist practice. Phys Ther. 2009 Mar;89(3):267-82. doi: 10.2522/ptj.20080130. Epub 2009 Jan 23. PMID 19168711
- [Background] Garre-Olmo J, Faundez-Zanuy M, Lopez-de-Ipina K, Calvo-Perxas L, Turro-Garriga O. Kinematic and Pressure Features of Handwriting and Drawing: Preliminary Results Between Patients with Mild Cognitive Impairment, Alzheimer Disease and Healthy Controls. Curr Alzheimer Res. 2017;14(9):960-968. doi: 10.2174/1567205014666170309120708. PMID 28290244
- [Background] Engel-Yeger B, Hus S, Rosenblum S. Age effects on sensory-processing abilities and their impact on handwriting. Can J Occup Ther. 2012 Dec;79(5):264-74. doi: 10.2182/CJOT.2012.79.5.2. PMID 23539771
- [Background] Dixon RA, Kurzman D, Friesen IC. Handwriting performance in younger and older adults: age, familiarity, and practice effects. Psychol Aging. 1993 Sep;8(3):360-70. doi: 10.1037//0882-7974.8.3.360. PMID 8216956
- See also: Neuroscript software — http://www.neuroscript.net/movalyzer.php
- See also: Movesense — http://www.movesense.com/wp-content/uploads/2023/04/Movesense-Medical-Instructions-For-Use-5.0-03-2023.pdf